CLINICAL TRIAL: NCT06882057
Title: Chinese Children's Cancer Group-2025 Protocol for Newly Diagnosed Low Risk Childhood B-cell Acute Lymphoblastic Leukemia
Brief Title: Newly-diagnosed Low Risk Pediatric B-cell ALL Protocol
Acronym: CCCG-LR-B-ALL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025021
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia ALL; Childhood Leukemia, Acute Lymphoblastic; B Cell Acute Lymphoblastic Leukemia (B-ALL)
Keywords: blinatumomab; chemo-light
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — blinatumomab; Dexamethasone; Prednisone; Asparaginase; Vincristine; Cytarabine; Methotrexate; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NGS MRD46 ≥ 10^-6 (Experimental): All LR-B-ALL patients will be treated with 14 days of blinatumomab (Blina-14) as early intensification to replace CAT+ (historically given in LR-B-AL with MRD19>0.1% in the 2020 protocol). Additionally, second 14 days of blinatumomab will be given after completion of HDMTX consolidation treatment. Reinduction-2 and Maintenance-2 will be given in full doses
  Interventions: Drug: Blinatumomab
- MRD19≥ 0.01% and NGS MRD46 < 10^-6 (Experimental): All LR-B-ALL patients will be treated with 14 days of blinatumomab (Blina-14) as early intensification to replace CAT+ (historically given in LR-B-AL with MRD19>0.1% in the 2020 protocol). Additionally, second 14 days of blinatumomab will be given after completion of HDMTX consolidation treatment. Reinduction-2 will be omitted, but Maintenance-2 will be given in full doses
- MRD19 < 0.01% and NGS MRD46 < 10^-6 (Experimental): All LR-B-ALL patients will be treated with 14 days of blinatumomab (Blina-14) as early intensification to replace CAT+ (historically given in LR-B-AL with MRD19>0.1% in the 2020 protocol). Additionally, second 14 days of blinatumomab will be given after completion of HDMTX consolidation treatment. Reinduction-2 will be omitted, and 5 cycles of Maintenance-2 will be omitted
  Interventions: Drug: Blinatumomab; Drug: Reinduction-2 omission; Drug: Chemo-light Maintenance 2

INTERVENTIONS:
Drug: Blinatumomab — All LR-B-ALL patients will be treated with 14 days of blinatumomab (Blina-14) as early intensification to replace CAT+ (historically given in LR-B-AL with MRD19>0.1% in the 2020 protocol). Additionally, second 14 days of blinatumomab will be given after completion of HDMTX consolidation treatment.
  Other Names: Dexamethasone; Prednisone; Asparaginase; Vincristine; Cyclophosphomide; Cytarabine; 6-MP; Methotrexate; Daunorubicin
  Arms: MRD19 < 0.01% and NGS MRD46 < 10^-6; NGS MRD46 ≥ 10^-6
Drug: Reinduction-2 omission — Reinduction-2 will be omitted for patients with NGS-MRD46<10^-6 who have receive the two courses of Blina-14.
  Other Names: Dexamethasone; Prednisone; Daunorubicin; Asparaginase; Vincristine; Cyclophosphomide; Cytarabine; 6-MP; Methotrexate
  Arms: MRD19 < 0.01% and NGS MRD46 < 10^-6
Drug: Chemo-light Maintenance 2 — Patients with FCM-MRD19<0.01% and IgH rearrangement NGS MRD 46<10^-6 will receive chemo-light maintenance-2 with 4 cyles of 8-week course of MTX + 6MP (totally 32 weeks).
  Other Names: Dexamethasone; Prednisone; Daunorubicin; Asparaginase; Vincristine; Cyclophosphomide; Cytarabine; 6-MP; Methotrexate
  Arms: MRD19 < 0.01% and NGS MRD46 < 10^-6

SUMMARY:
CCCG-ALL2025 LR-B-ALL plan is designed based on the CCCG-ALL2020 plan. This is a clinical trial using 14 days of blinatumomab (Blina-14) as early intensification after induction therapy and 2nd Blina-14 in consolidation therapy in all newly diagnosed provisional low-risk (LR) pediatric acute lymphoblastic leukemia (ALL) patients, regardless of measurable residual diseases (MRD) status. We will compare the efficacy of chemotherapy combined with Blina-14, comparing to CAT+ intensification or historical regimens. Patients with early remission in depth will receive chemo-light late intensification and maintenance therapy afterwards. Early complete remission in depth and maintenance reduction will be determined by next-generation sequencing (Ig-NGS MRD).

DETAILED DESCRIPTION:
1. All LR-B-ALL patients will be treated with 14 days of blinatumomab (Blina-14) as early intensification to replace CAT+ (historically given in LR-B-AL with MRD19>0.1% in the 2020 protocol).
2. Two courses of HD-MTX will be administered as consolidation phase, maintaining the same dose of 3 g/m².
3. Second 14 days of blinatumomab will be given after completion of HDMTX consolidation treatment .
4. Adding IgH rearrangement NGS MRD as an evaluation indicator. Reinduction-2 will be omitted for patients with NGS-MRD46<10-6 who have receive the second course of Blina-14. (Reinduction-2 should be given regardless of NGS-MRD 46 status in patients who did not receive the second course of binatumomab).
5. A total of four repeating courses will be applied in Maintenance 1 (in contrast to 5 courses in 2020 protocol). Additionally, one-week rest period will be implemented after each course to ensure safety and optimal efficacy.
6. Patients with FCM-MRD19<0.01% and IgH rearrangement NGS MRD 46<10-6 will receive chemo-light maintenance-2 with 4 cyles of 8-week course of MTX + 6MP (totally 32 weeks). The other patients with higher levels of MRD by FCM MRD or NGS MRD will receive maintenance-2 with 9 cycles of 8-week course of MTX + 6MP for a total of 72 weeks (same as CCCG-ALL2020)
7. Bone Marrow Aspiration Assessment (BMA): One additional bone marrow puncture at the end of 1st Blina-14 course (Day60 MRD) will be performed at early intensification phase. This results in a total of 4 BMAs in the CCCG2025-LR protocol, in contrast to 3 BMAs in 2020 protocol.
8. Triple Intrathecal Therapy (TIT)：In the HDMTX consolidation phase, there will be two TITs in contrast to four treatments in the CCCG2020 protocol. To compensate for this reduction, two additional TIT treatments will be administrated before the 1st and 2nd Blina-14 courses. Additionally, two intrathecal treatments will be added during Reinduction 1 and Reinduction 2 to further enhance CNS control. Meanwhile, one TIT will be reduced in the Maintenance-1 phase compared to 2020 protocol. This results in a total of 16 or 17 TITs, depending on whether the second Blina-14 course is applied This is similar to the CCCG2020, where 16 or 17 TITs are administrated depending on whether CAT+ was given).
9. Adding pharmacotyping study for LR B-ALL.
10. Treatment duration: The treatment duration for the CCCG-LR-ALL-2020 protocol is 121/124 weeks (depending on if CAT+ was given). In the CCCG-LR-ALL-2025 protocol:

    * For patients with NGS MRD46 ≥10-6, the total treatment duration is 123 weeks. Key changes include: 2 weeks of Blina-14 replacing 3 weeks of CAT+, 2 courses of HDMTX reduction (4 weeks), and an additional 2 weeks for the 2nd blina-14 course added following HDMTX;
    * For patients with MRD19≥ 0.01% and NGS MRD46 < 10-6 who subsequently receive 2nd Blina-14, Reinduction-2 is omitted, shortening the total duration by 3 weeks. (120 weeks in total). If the 2nd Blina-14 is not administrated, Reinduction -2 will still be included, resulting in a total duration of 121 weeks.
    * For patients with MRD19 < 0.01% and NGS MRD46 < 10-6, who subsequently receive 2nd Blina-14, both the Reinduction-2 (3 weeks) and the subsequent 5 cycles of Maintenance-2 (40 weeks) are omitted. This results in a total treatment duration of 80 weeks (81 weeks if 2nd Blina-14 is not applied).

ELIGIBILITY:
Inclusion Criteria:

Must meet all items below:

1. Age older than 1 year and younger than 18 years.
2. Diagnosis of acute lymphoblastic leukemia by bone marrow morphology.
3. Diagnosis of B-ALL by immunophenotyping.
4. Low risk group

Exclusion Criteria:

Should be excluded in the presence of any item below:

1. T-ALL
2. I/HR B-ALL group
3. sIgM+
4. Acute leukemias of ambiguous lineage diagnosed according to WHO or EGIL criteria.
5. Philadelphia chromosome positive ALL (Ph-ALL)
6. ALL evolved from chronic myeloid leukemia (CML).
7. Down's syndrome, or major congenital or hereditary disease with organ dysfunction
8. Secondary leukemia
9. Known underlying congenital immunodeficiency or metabolic disease
10. Congenital heart disease with cardiac insufficiency.
11. Glucocorticoid treatment for ≥14 days, or ABL kinase inhibitors for > 7 days within one month before enrollment, or any chemotherapy or radiotherapy within 3 months before enrollment (except for emergency radiotherapy to relieve airway compression)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Compare 3-year event-free survival (EFS) between patients who receive Blina-14 intensification with this historical controls from CCCG-ALL2015 and CCCG-ALL2000 | The expected study duration is approximately 5 years.
  The primary historical control cohort consists of the patients on the CCCG-ALL2020 trial determined as LR after remission indiction, received 2xHDMTX during consolidation and did not receive Bliniatumomab. As of end of 2024, this cohort contains 1111 patients, with 3-year EFS 0.963 and standard error 0.0087, 95% confidence interval [0.953,0.980] . The sample size and power assessment below is based on these data.
  The primary comparison is between the patients on this trial who are determined as LR after remission induction to the historical cohort described above, on 3-year EFS probability.
  .Power of the above test procedure is assessed by a simulation study. Historical control is set from the preliminary data as S0=0.963,v0^2=0.0087^2. For the current trial total sample size is set to n=2325 with 5 year accrual.LN distribution is chosen for its good assemblance of the EFS functions of the LR cohorts in the historical data.

SECONDARY OUTCOMES:
Estimate event-free survival (EFS) in patients with deep remission (FCM MRD19<0.01% and Ig-NGS MRD46<10-6) who received Maintenance-2' with reduced intensity chemotherapy | Approximately 6.5 years.
  The EFS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 1, 3, 5 years since diagnosis).
Estimate overall survival (OS) in patients with deep remission (FCM MRD19<0.01% and Ig-NGS MRD46<10-6) who received Maintenance-2' with reduced intensity chemotherapy | Approximately 6.5 years.
  The OS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 1, 3, 5 years since diagnosis).
Estimate cumulative incidence of relapse (CIR) in patients with deep remission (FCM MRD19<0.01% and Ig-NGS MRD46<10-6) who received Maintenance-2' with reduced intensity chemotherapy | Approximately 6.5 years.
  The CIR curve will be estimated by Kalbafleisch-Prentice method, along with 95% confidence intervals.
Compare event-free survival (EFS) to those of historical cohorts (CCCG-ALL-2015 and CCCG-ALL2020) | Approximately 6.5 years.
  The EFS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 1, 3, 5 years since diagnosis). Standard error will be estimated using the default procedure in R. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of EFS will be performed using two-sided log-rank test. Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
Compare overall survival (OS) to those of historical cohorts (CCCG-ALL-2015 and CCCG-ALL2020) | Approximately 6.5 years.
  The OS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 1, 3, 5 years since diagnosis). Comparison of OS functions will be conducted using the two-sided log-rank test. Standard error will be estimated using the default procedure in R. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of OS will be performed using two-sided log-rank test. Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
Compare cumulative incidence of relapse (CIR) to those of historical cohorts (CCCG-ALL-2015 and CCCG-ALL2020) | Approximately 6.5 years.
  CIR functions of relapse will be estimated by the Kalbafleisch-Prentice method. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of CIR will be performed by Gray's test. Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Fine-Gray models.
Compare event-free survival (EFS) between patients with deepen remission (FCM MRD19<0.01% and Ig-NGS MRD46<10-6) who receive one course of Blina-14 and those who recevive two courses of Blina-14. | Approximately 6.5 years
  The EFS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 1, 3, 5 years since diagnosis). Standard error will be estimated using the default procedure in R. Comparisons of EFS will be performed using two-sided log-rank test. Multivariable regression modeling including known prognostic factors as main effects may also be performed, using the Cox models.
Compare overall survival (OS) between patients with deepen remission (FCM MRD19<0.01% and Ig-NGS MRD46<10-6) who receive one course of Blina-14 and those who recevive two courses of Blina-14. | Approximately 6.5 years
  The OS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 1, 3, 5 years since diagnosis). Standard error will be estimated using the default procedure in R. Comparisons of OS will be performed using two-sided log-rank test. Multivariable regression modeling including known prognostic factors as main effects may also be performed, using the Cox models.
Compare cumulative incidence of relapse (CIR) between patients with deepen remission (FCM MRD19<0.01% and Ig-NGS MRD46<10-6) who receive one course of Blina-14 and those who recevive two courses of Blina-14. | Approximately 6.5 years
  CIR functions of relapse will be estimated by the Kalbafleisch-Prentice method. Comparisons of CIR will be performed by Gray's test. Multivariable regression modeling including known prognostic factors as main effects may also be performed, using the Fine-Gray models.

OTHER OUTCOMES:
Compare the 3-year EFS between patients who received Blina-14 intensification with those who received CAT+ intensification | Approximately 3.5 years
  The EFS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at 3 years since diagnosis. Standard error will be estimated using the default procedure in R. Comparison will be made using the Z-test procedure described in primary endpoint.
Evaluate the significance of the early deep remission rate after Blina-14 intensification by its association with treatment outcomes, especially cumulative incidence of relapse (CIR) | Approximately 6.5 years.
  CIR functions of relapse will be estimated by the Kalbafleisch-Prentice method. Associations between deep remission status after blinatumimab treatment and relapse will be analysed using Gray's test or Fine-Gray regression models, as appropriate.
Evaluate toxicities during the immuno-chemo combined therapy in provisional LR-ALL. | Up to 30 days after last dose of study treatment
  Proportions of grade-3 or higher AEs in each treatment phase will be estimated by the sample proportions along with exact 95% confidence intervals. Cumulative incidences of various grade-3 or higher AEs throughout therapy will be estimated by the Kalbafleisch-Prentice method; death, relapse and other events rendering off therapy before completion are regarded as competing risks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, MD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, CAMS & PUMC
Locations (27):
- China (26):
  - Anhui Medical University Second Affiliated Hospital, Hefei, Anhui
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Chongqing Medical University Affiliated Children's Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Children's Hospital, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of the Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Nanjing Children's Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Children's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Children's Medical Cener, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Xi'an Northwest Women and Children Hospital, Xi’an, Shanxi
  - Shenzhen Children's Hospita, Shenzhen, Shenzhen
  - West China Second University Hospital, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, CAMS & PUMC, Tianjin, Tianjin Municipality
- Hong Kong Children's Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
1. Demographic Data: Age, sex, and other relevant baseline characteristics.
  2. Treatment Information: Data on interventions received by participants, including dosage, treatment cycles, and duration.
  3. Outcome Measures: Detailed information on primary and secondary outcome measures, such as response rates, survival rates, adverse events, and any the pre-specified endpoints.
  4. Adverse Events: Data on all reported adverse events, including severity, duration, and outcome.
  5. Laboratory Data: Results from laboratory tests, such as blood counts, biochemical markers, or molecular analysis.
  6. Medical History: Pre-existing conditions, comorbidities, and prior treatments or interventions.
  7. Vital Signs: relevant physiological data.
  8. Efficacy and Safety Data: Any data relating to the efficacy (e.g., event-free survival) and safety (e.g., adverse effects) of the treatment.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available upon publication of the primary trial results or after trial completion, whichever occurs first, starting on 2032, and will remain accessible for 5 years.
Access Criteria: Researchers, healthcare professionals who meet the criteria for access (e.g., academic researchers conducting secondary analyses or regulatory bodies reviewing safety data) will be able to request access to de-identified IPD and supporting information. Access will be facilitated through clinical trials.gov/emailing to PI, where users can submit a request and provide a research proposal. Data access will be granted after a formal review and approval process, subject to compliance with the data-sharing agreement and confidentiality terms.
URL: http://cccg.nipher.com/cccg/

REFERENCES:
- [Background] Lee SHR, Yang W, Gocho Y, John A, Rowland L, Smart B, Williams H, Maxwell D, Hunt J, Yang W, Crews KR, Roberts KG, Jeha S, Cheng C, Karol SE, Relling MV, Rosner GL, Inaba H, Mullighan CG, Pui CH, Evans WE, Yang JJ. Pharmacotypes across the genomic landscape of pediatric acute lymphoblastic leukemia and impact on treatment response. Nat Med. 2023 Jan;29(1):170-179. doi: 10.1038/s41591-022-02112-7. Epub 2023 Jan 5. PMID 36604538
- [Background] Chen H, Gu M, Liang J, Song H, Zhang J, Xu W, Zhao F, Shen D, Shen H, Liao C, Tang Y, Xu X. Minimal residual disease detection by next-generation sequencing of different immunoglobulin gene rearrangements in pediatric B-ALL. Nat Commun. 2023 Nov 17;14(1):7468. doi: 10.1038/s41467-023-43171-9. PMID 37978187
- [Background] Hengeveld PJ, van der Klift MY, Kolijn PM, Davi F, Kavelaars FG, de Jonge E, Robrecht S, Assmann JLJC, van der Straten L, Ritgen M, Westerweel PE, Fischer K, Goede V, Hallek M, Levin MD, Langerak AW. Detecting measurable residual disease beyond 10-4 by an IGHV leader-based NGS approach improves prognostic stratification in CLL. Blood. 2023 Feb 2;141(5):519-528. doi: 10.1182/blood.2022017411. PMID 36084320
- [Background] Svaton M, Skotnicova A, Reznickova L, Rennerova A, Valova T, Kotrova M, van der Velden VHJ, Bruggemann M, Darzentas N, Langerak AW, Zuna J, Stary J, Trka J, Fronkova E. NGS better discriminates true MRD positivity for the risk stratification of childhood ALL treated on an MRD-based protocol. Blood. 2023 Feb 2;141(5):529-533. doi: 10.1182/blood.2022017003. PMID 36240445
- [Background] Li Z, Jiang N, Lim EH, Chin WHN, Lu Y, Chiew KH, Kham SKY, Yang W, Quah TC, Lin HP, Tan AM, Ariffin H, Yang JJ, Yeoh AE. Identifying IGH disease clones for MRD monitoring in childhood B-cell acute lymphoblastic leukemia using RNA-Seq. Leukemia. 2020 Sep;34(9):2418-2429. doi: 10.1038/s41375-020-0774-4. Epub 2020 Feb 25. PMID 32099036
- [Background] Foa R, Bassan R, Elia L, Piciocchi A, Soddu S, Messina M, Ferrara F, Lunghi M, Mule A, Bonifacio M, Fracchiolla N, Salutari P, Fazi P, Guarini A, Rambaldi A, Chiaretti S. Long-Term Results of the Dasatinib-Blinatumomab Protocol for Adult Philadelphia-Positive ALL. J Clin Oncol. 2024 Mar 10;42(8):881-885. doi: 10.1200/JCO.23.01075. Epub 2023 Dec 21. PMID 38127722
- [Background] Hogan LE, Brown PA, Ji L, Xu X, Devidas M, Bhatla T, Borowitz MJ, Raetz EA, Carroll A, Heerema NA, Zugmaier G, Sharon E, Bernhardt MB, Terezakis SA, Gore L, Whitlock JA, Hunger SP, Loh ML. Children's Oncology Group AALL1331: Phase III Trial of Blinatumomab in Children, Adolescents, and Young Adults With Low-Risk B-Cell ALL in First Relapse. J Clin Oncol. 2023 Sep 1;41(25):4118-4129. doi: 10.1200/JCO.22.02200. Epub 2023 May 31. PMID 37257143
- [Background] Litzow MR, Sun Z, Mattison RJ, Paietta EM, Roberts KG, Zhang Y, Racevskis J, Lazarus HM, Rowe JM, Arber DA, Wieduwilt MJ, Liedtke M, Bergeron J, Wood BL, Zhao Y, Wu G, Chang TC, Zhang W, Pratz KW, Dinner SN, Frey N, Gore SD, Bhatnagar B, Atallah EL, Uy GL, Jeyakumar D, Lin TL, Willman CL, DeAngelo DJ, Patel SB, Elliott MA, Advani AS, Tzachanis D, Vachhani P, Bhave RR, Sharon E, Little RF, Erba HP, Stone RM, Luger SM, Mullighan CG, Tallman MS. Blinatumomab for MRD-Negative Acute Lymphoblastic Leukemia in Adults. N Engl J Med. 2024 Jul 25;391(4):320-333. doi: 10.1056/NEJMoa2312948. PMID 39047240
- [Background] van der Sluis IM, de Lorenzo P, Kotecha RS, Attarbaschi A, Escherich G, Nysom K, Stary J, Ferster A, Brethon B, Locatelli F, Schrappe M, Scholte-van Houtem PE, Valsecchi MG, Pieters R. Blinatumomab Added to Chemotherapy in Infant Lymphoblastic Leukemia. N Engl J Med. 2023 Apr 27;388(17):1572-1581. doi: 10.1056/NEJMoa2214171. PMID 37099340
- [Background] Foa R, Bassan R, Vitale A, Elia L, Piciocchi A, Puzzolo MC, Canichella M, Viero P, Ferrara F, Lunghi M, Fabbiano F, Bonifacio M, Fracchiolla N, Di Bartolomeo P, Mancino A, De Propris MS, Vignetti M, Guarini A, Rambaldi A, Chiaretti S; GIMEMA Investigators. Dasatinib-Blinatumomab for Ph-Positive Acute Lymphoblastic Leukemia in Adults. N Engl J Med. 2020 Oct 22;383(17):1613-1623. doi: 10.1056/NEJMoa2016272. PMID 33085860
- [Background] Gupta S, Rau RE, Kairalla JA, Rabin KR, Wang C, Angiolillo AL, Alexander S, Carroll AJ, Conway S, Gore L, Kirsch I, Kubaney HR, Li AM, McNeer JL, Militano O, Miller TP, Moyer Y, O'Brien MM, Okada M, Reshmi SC, Shago M, Wagner E, Winick N, Wood BL, Haworth-Wright T, Zaman F, Zugmaier G, Zupanec S, Devidas M, Hunger SP, Teachey DT, Raetz EA, Loh ML. Blinatumomab in Standard-Risk B-Cell Acute Lymphoblastic Leukemia in Children. N Engl J Med. 2025 Feb 27;392(9):875-891. doi: 10.1056/NEJMoa2411680. Epub 2024 Dec 7. PMID 39651791
- [Background] Kantarjian H, Stein A, Gokbuget N, Fielding AK, Schuh AC, Ribera JM, Wei A, Dombret H, Foa R, Bassan R, Arslan O, Sanz MA, Bergeron J, Demirkan F, Lech-Maranda E, Rambaldi A, Thomas X, Horst HA, Bruggemann M, Klapper W, Wood BL, Fleishman A, Nagorsen D, Holland C, Zimmerman Z, Topp MS. Blinatumomab versus Chemotherapy for Advanced Acute Lymphoblastic Leukemia. N Engl J Med. 2017 Mar 2;376(9):836-847. doi: 10.1056/NEJMoa1609783. PMID 28249141
- [Background] von Stackelberg A, Locatelli F, Zugmaier G, Handgretinger R, Trippett TM, Rizzari C, Bader P, O'Brien MM, Brethon B, Bhojwani D, Schlegel PG, Borkhardt A, Rheingold SR, Cooper TM, Zwaan CM, Barnette P, Messina C, Michel G, DuBois SG, Hu K, Zhu M, Whitlock JA, Gore L. Phase I/Phase II Study of Blinatumomab in Pediatric Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia. J Clin Oncol. 2016 Dec 20;34(36):4381-4389. doi: 10.1200/JCO.2016.67.3301. Epub 2016 Oct 31. PMID 27998223
- [Background] Topp MS, Gokbuget N, Stein AS, Zugmaier G, O'Brien S, Bargou RC, Dombret H, Fielding AK, Heffner L, Larson RA, Neumann S, Foa R, Litzow M, Ribera JM, Rambaldi A, Schiller G, Bruggemann M, Horst HA, Holland C, Jia C, Maniar T, Huber B, Nagorsen D, Forman SJ, Kantarjian HM. Safety and activity of blinatumomab for adult patients with relapsed or refractory B-precursor acute lymphoblastic leukaemia: a multicentre, single-arm, phase 2 study. Lancet Oncol. 2015 Jan;16(1):57-66. doi: 10.1016/S1470-2045(14)71170-2. Epub 2014 Dec 16. PMID 25524800
- [Background] Brown PA, Ji L, Xu X, Devidas M, Hogan LE, Borowitz MJ, Raetz EA, Zugmaier G, Sharon E, Bernhardt MB, Terezakis SA, Gore L, Whitlock JA, Pulsipher MA, Hunger SP, Loh ML. Effect of Postreinduction Therapy Consolidation With Blinatumomab vs Chemotherapy on Disease-Free Survival in Children, Adolescents, and Young Adults With First Relapse of B-Cell Acute Lymphoblastic Leukemia: A Randomized Clinical Trial. JAMA. 2021 Mar 2;325(9):833-842. doi: 10.1001/jama.2021.0669. PMID 33651090
- [Background] Mattano LA Jr, Devidas M, Maloney KW, Wang C, Friedmann AM, Buckley P, Borowitz MJ, Carroll AJ, Gastier-Foster JM, Heerema NA, Kadan-Lottick NS, Matloub YH, Marshall DT, Stork LC, Loh ML, Raetz EA, Wood BL, Hunger SP, Carroll WL, Winick NJ. Favorable Trisomies and ETV6-RUNX1 Predict Cure in Low-Risk B-Cell Acute Lymphoblastic Leukemia: Results From Children's Oncology Group Trial AALL0331. J Clin Oncol. 2021 May 10;39(14):1540-1552. doi: 10.1200/JCO.20.02370. Epub 2021 Mar 19. PMID 33739852
- [Background] Campbell M, Kiss C, Zimmermann M, Riccheri C, Kowalczyk J, Felice MS, Kuzmanovic M, Kovacs G, Kosmidis H, Gonzalez A, Bilic E, Castillo L, Kolenova A, Jazbec J, Popa A, Konstantinov D, Kappelmayer J, Szczepanski T, Dworzak M, Buldini B, Gaipa G, Marinov N, Rossi J, Nagy A, Gaspar I, Stary J, Schrappe M. Childhood Acute Lymphoblastic Leukemia: Results of the Randomized Acute Lymphoblastic Leukemia Intercontinental-Berlin-Frankfurt-Munster 2009 Trial. J Clin Oncol. 2023 Jul 1;41(19):3499-3511. doi: 10.1200/JCO.22.01760. Epub 2023 May 4. PMID 37141547
- [Background] Aldoss I, Song J, Stiller T, Nguyen T, Palmer J, O'Donnell M, Stein AS, Marcucci G, Forman S, Pullarkat V. Correlates of resistance and relapse during blinatumomab therapy for relapsed/refractory acute lymphoblastic leukemia. Am J Hematol. 2017 Sep;92(9):858-865. doi: 10.1002/ajh.24783. Epub 2017 Jun 5. PMID 28494518
- [Background] Kantarjian HM, DeAngelo DJ, Advani AS, Stelljes M, Kebriaei P, Cassaday RD, Merchant AA, Fujishima N, Uchida T, Calbacho M, Ejduk AA, O'Brien SM, Jabbour EJ, Zhang H, Sleight BJ, Vandendries ER, Marks DI. Hepatic adverse event profile of inotuzumab ozogamicin in adult patients with relapsed or refractory acute lymphoblastic leukaemia: results from the open-label, randomised, phase 3 INO-VATE study. Lancet Haematol. 2017 Aug;4(8):e387-e398. doi: 10.1016/S2352-3026(17)30103-5. Epub 2017 Jul 4. PMID 28687420
- [Background] Orlando EJ, Han X, Tribouley C, Wood PA, Leary RJ, Riester M, Levine JE, Qayed M, Grupp SA, Boyer M, De Moerloose B, Nemecek ER, Bittencourt H, Hiramatsu H, Buechner J, Davies SM, Verneris MR, Nguyen K, Brogdon JL, Bitter H, Morrissey M, Pierog P, Pantano S, Engelman JA, Winckler W. Genetic mechanisms of target antigen loss in CAR19 therapy of acute lymphoblastic leukemia. Nat Med. 2018 Oct;24(10):1504-1506. doi: 10.1038/s41591-018-0146-z. Epub 2018 Oct 1. PMID 30275569
- [Background] Cordoba S, Onuoha S, Thomas S, Pignataro DS, Hough R, Ghorashian S, Vora A, Bonney D, Veys P, Rao K, Lucchini G, Chiesa R, Chu J, Clark L, Fung MM, Smith K, Peticone C, Al-Hajj M, Baldan V, Ferrari M, Srivastava S, Jha R, Arce Vargas F, Duffy K, Day W, Virgo P, Wheeler L, Hancock J, Farzaneh F, Domning S, Zhang Y, Khokhar NZ, Peddareddigari VGR, Wynn R, Pule M, Amrolia PJ. CAR T cells with dual targeting of CD19 and CD22 in pediatric and young adult patients with relapsed or refractory B cell acute lymphoblastic leukemia: a phase 1 trial. Nat Med. 2021 Oct;27(10):1797-1805. doi: 10.1038/s41591-021-01497-1. Epub 2021 Oct 12. PMID 34642489
- [Background] Ruella M, Korell F, Porazzi P, Maus MV. Mechanisms of resistance to chimeric antigen receptor-T cells in haematological malignancies. Nat Rev Drug Discov. 2023 Dec;22(12):976-995. doi: 10.1038/s41573-023-00807-1. Epub 2023 Oct 31. PMID 37907724
- [Background] Leung KT, Cai J, Liu Y, Chan KYY, Shao J, Yang H, Hu Q, Xue Y, Wu X, Guo X, Zhai X, Wang N, Li X, Tian X, Li Z, Xue N, Guo Y, Wang L, Zou Y, Xiao P, He Y, Jin R, Tang J, Yang JJ, Shen S, Pui CH, Li CK. Prognostic implications of CD9 in childhood acute lymphoblastic leukemia: insights from a nationwide multicenter study in China. Leukemia. 2024 Feb;38(2):250-257. doi: 10.1038/s41375-023-02089-3. Epub 2023 Nov 25. PMID 38001171
- [Background] Li B, Brady SW, Ma X, Shen S, Zhang Y, Li Y, Szlachta K, Dong L, Liu Y, Yang F, Wang N, Flasch DA, Myers MA, Mulder HL, Ding L, Liu Y, Tian L, Hagiwara K, Xu K, Zhou X, Sioson E, Wang T, Yang L, Zhao J, Zhang H, Shao Y, Sun H, Sun L, Cai J, Sun HY, Lin TN, Du L, Li H, Rusch M, Edmonson MN, Easton J, Zhu X, Zhang J, Cheng C, Raphael BJ, Tang J, Downing JR, Alexandrov LB, Zhou BS, Pui CH, Yang JJ, Zhang J. Therapy-induced mutations drive the genomic landscape of relapsed acute lymphoblastic leukemia. Blood. 2020 Jan 2;135(1):41-55. doi: 10.1182/blood.2019002220. PMID 31697823
- [Background] Brady SW, Roberts KG, Gu Z, Shi L, Pounds S, Pei D, Cheng C, Dai Y, Devidas M, Qu C, Hill AN, Payne-Turner D, Ma X, Iacobucci I, Baviskar P, Wei L, Arunachalam S, Hagiwara K, Liu Y, Flasch DA, Liu Y, Parker M, Chen X, Elsayed AH, Pathak O, Li Y, Fan Y, Michael JR, Rusch M, Wilkinson MR, Foy S, Hedges DJ, Newman S, Zhou X, Wang J, Reilly C, Sioson E, Rice SV, Pastor Loyola V, Wu G, Rampersaud E, Reshmi SC, Gastier-Foster J, Guidry Auvil JM, Gesuwan P, Smith MA, Winick N, Carroll AJ, Heerema NA, Harvey RC, Willman CL, Larsen E, Raetz EA, Borowitz MJ, Wood BL, Carroll WL, Zweidler-McKay PA, Rabin KR, Mattano LA, Maloney KW, Winter SS, Burke MJ, Salzer W, Dunsmore KP, Angiolillo AL, Crews KR, Downing JR, Jeha S, Pui CH, Evans WE, Yang JJ, Relling MV, Gerhard DS, Loh ML, Hunger SP, Zhang J, Mullighan CG. The genomic landscape of pediatric acute lymphoblastic leukemia. Nat Genet. 2022 Sep;54(9):1376-1389. doi: 10.1038/s41588-022-01159-z. Epub 2022 Sep 1. PMID 36050548
- [Background] Newman S, Nakitandwe J, Kesserwan CA, Azzato EM, Wheeler DA, Rusch M, Shurtleff S, Hedges DJ, Hamilton KV, Foy SG, Edmonson MN, Thrasher A, Bahrami A, Orr BA, Klco JM, Gu J, Harrison LW, Wang L, Clay MR, Ouma A, Silkov A, Liu Y, Zhang Z, Liu Y, Brady SW, Zhou X, Chang TC, Pande M, Davis E, Becksfort J, Patel A, Wilkinson MR, Rahbarinia D, Kubal M, Maciaszek JL, Pastor V, Knight J, Gout AM, Wang J, Gu Z, Mullighan CG, McGee RB, Quinn EA, Nuccio R, Mostafavi R, Gerhardt EL, Taylor LM, Valdez JM, Hines-Dowell SJ, Pappo AS, Robinson G, Johnson LM, Pui CH, Ellison DW, Downing JR, Zhang J, Nichols KE. Genomes for Kids: The Scope of Pathogenic Mutations in Pediatric Cancer Revealed by Comprehensive DNA and RNA Sequencing. Cancer Discov. 2021 Dec 1;11(12):3008-3027. doi: 10.1158/2159-8290.CD-20-1631. PMID 34301788
- [Background] Teachey DT, Pui CH. Comparative features and outcomes between paediatric T-cell and B-cell acute lymphoblastic leukaemia. Lancet Oncol. 2019 Mar;20(3):e142-e154. doi: 10.1016/S1470-2045(19)30031-2. PMID 30842058
- [Background] Jeha S, Pei D, Choi J, Cheng C, Sandlund JT, Coustan-Smith E, Campana D, Inaba H, Rubnitz JE, Ribeiro RC, Gruber TA, Raimondi SC, Khan RB, Yang JJ, Mullighan CG, Downing JR, Evans WE, Relling MV, Pui CH. Improved CNS Control of Childhood Acute Lymphoblastic Leukemia Without Cranial Irradiation: St Jude Total Therapy Study 16. J Clin Oncol. 2019 Dec 10;37(35):3377-3391. doi: 10.1200/JCO.19.01692. Epub 2019 Oct 28. PMID 31657981
- See also: CCCG-ALL-2025 DATASET — http://cccg.nipher.com/cccg/
- Available data/document: Individual Participant Data Set: CCCG-ALL — http://cccg.nipher.com/cccg/ — CCCG-ALL-2025 DATASET